CLINICAL TRIAL: NCT07171515
Title: Development & Clinical Application of K-PaC Registry Version 2.0
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang Myung Woo, Head, Center for Liver and Pancreatobiliary Cancer, National Cancer Center, Korea
Other Study IDs: NCC2022-0061
Record Dates: First submitted 2025-06-15; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Transcriptome, Whole genome, Epigenome, Proteome, Metabolome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development and clinical use of pancreatic cancer registry

* Development of K-PaC Registry v.2.0: Retrospective data integration from 2010 to 2022 and prospective data collection from more than 811 enrolled patients from 2023 to 2029
* Creation of clinical evidence (RWE) based on pancreatic cancer real-world data (RWD): 3 or more

DETAILED DESCRIPTION:
We plan to collect retrospective and prospective data based on medical data centered on EMR. ∙ This registry is built on EMR data containing specific information on medical provider records and patient health records. It is designed to enable the confirmation of specific treatment history and medical staff records, and to generate highly valid RWD-based evidence through EMR information such as accurate diagnosis of disease, treatment method, symptom changes, monitoring of lab data values, and patient status. ∙ Based on the built registry data, it is possible to conduct research based on evaluation of drug treatment and additional comparison of indications for elderly or poor general condition patients who are excluded from regular clinical trials, as well as research on diagnosis and prognosis. The clinical information and biomarkers of the prospective patient group are analyzed to evaluate the correlation with treatment response, overall and progression-free survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pancreatic cancer

Exclusion Criteria:

* In cases where medical record review is not feasible

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 6923 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and clinical use of a pancreatic cancer registry | From initial diagnosis to death
  Development of K-PaC Registry v.2.0: Retrospective data integration from 2010 to 2022 and prospective data collection from more than 811 enrolled patients from 2023 to 2029Creation of clinical evidence (RWE) based on pancreatic cancer real-world data (RWD): 3 or more

SECONDARY OUTCOMES:
Assessing the association between pancreatic cancer biomarker markers and treatment response, overall and progression-free survival | From initial diagnosis to death
  Transcriptome, Whole genome, Epigenome, Proteome, Metabolome

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No
There are restrictions under Korea's Personal Information Protection Act.

REFERENCES:
- See also: 1. Guidelines for the Pancreatic Cancer Registry, National Cancer Center Big Data Center — https://data.doi.or.kr/10.22694/CANCERDATA032018070101
- See also: 2. CONNECT Cancer Big Data Library: Pancreatic Cancer Section — https://cancerportal.kr/ncc/clinicalLibraryInfo.do
- See also: Korean clinical practice guideline for pancreatic cancer 2021: A summary of evidence-based, multi-disciplinary diagnostic and therapeutic approaches — https://www.kahbps.or.kr/bbs/index.kin?bbs_mode=view&f_wbcode=board_request&f_master_idx=770&f_template_type=list
- Available data/document: Study Protocol — https://data.doi.or.kr/10.22694/CANCERDATA032018070101 — 1. 1. Guidelines for the Pancreatic Cancer Registry, National Cancer Center Big Data
- Available data/document: Study Protocol — https://cancerportal.kr/ncc/clinicalLibraryInfo.do — 2. CONNECT Cancer Big Data Library: Pancreatic Cancer Section
- Available data/document: Study Protocol — https://www.kahbps.or.kr/bbs/index.kin?bbs_mode=view&f_wbcode=board_request&f_master_idx=770&f_template_type=list — Korean clinical practice guideline for pancreatic cancer 2021